CLINICAL TRIAL: NCT01246037
Title: Beta-blocker Therapy in Idiopathic Pulmonary Arterial Hypertension
Brief Title: Beta-blockers in i-PAH
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, A. Vonk Noordegraaf, Prof. dr., Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010-262
Record Dates: First submitted 2010-11-18; First posted 2010-11-23 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Idiopathic Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension; Beta-blocker; Adrenergic Receptor Antagonist
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension; Pulmonary Arterial Hypertension | interventions — Bisoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- First placebo (Experimental): First half year placebo, second half year bisoprolol
  Interventions: Drug: Bisoprolol
- First Bisoprolol (Experimental): First half year bisoprolol, second half year placebo
  Interventions: Drug: Bisoprolol

INTERVENTIONS:
Drug: Bisoprolol — In the first 4 months of study, the dose of the drug will be gradually increased; the titration scheme is based on the 'farmacotherapeutisch kompas' and monitored according to the ACC/AHA/ESC guidelines. Up titration will be performed under the responsibilities of an experienced heart failure cardiologist and pulmonologist.

SUMMARY:
The main question of this study is: 'Is selective beta-blocker treatment safe and effective in reducing sympathetic overdrive, thereby improving RV function and remodeling in patients with iPAH?'.

In addition to the determination of RVEF, the investigators will explore how beta-blocker therapy affects sympathetic overdrive, remodeling of the RV, single beat elastance, exercise capacity and mechanical efficiency.

30 iPAH patients will be randomized to either Bisoprolol- or placebo-treatment in a double-blinded fashion. A cross-over trial design will be used to increase the power of the study and to assess long-term effects of Bisoprolol-treatment and -withdrawal. The medication will be given in an escalating dose regimen (as described in the 'farmacotherapeutisch kompas', www.fk.cvz.nl) and treatment will be monitored along the guidelines of the American Heart Association.

DETAILED DESCRIPTION:
This is a clinical study aimed to provide a proof of concept of the safety and efficacy of beta-blocker treatment in PAH-associated right ventricular failure.

The protocol of the proposed double blinded cross over design.

The reasons for not choosing an initial open phase 1 study, but to start directly with a placebo controlled study are:

1. Although the drug is considered contraindicated in the studied patient population, it is very common for PAH patients to receive beta-blocker therapy in an uncontrolled way; without reports of serious side effects until now
2. Dose titration in the study will be performed on the basis of side-effects and at this moment the investigators cannot predict the optimal dose which is both safe and efficacious. Therefore, safety assessment can only be performed in combination with the assessment of pharmaceutical effectiveness.

After obtaining informed consent, 30 idiopathic PAH patients (NYHA II-III) will be randomly assigned to either the placebo group or beta-blocker therapy. For the randomization and study blinding the investigators will use a VUMC computer based procedure in close collaboration with the VUMC pharmacy.

In the first 4 months of study, the dose of the drug will be gradually increased; the titration scheme is based on the 'farmacotherapeutisch kompas' (described below) and monitored according to the ACC/AHA/ESC guidelines. Up titration will be performed under the responsibilities of an experienced heart failure cardiologist and pulmonologist.

MEASUREMENTS Time points 1, 3 and 5 (6 months periods): this includes a complete assessment of the patient

* Clinical assessment: physical examination, NYHA class, ECG, routine lab including NT-proBNP and urine tests for proteinuria.
* Imaging of right ventricular function: the primary measure of this study will be right ventricular ejection fraction measured by means of MRI. Additional MRI and echocardiographic measurements will be performed. (the complete study protocols are added as supplements).
* Right Heart Catheterization (performed under local anesthesia): Measurements of pressures in the pulmonary artery, right ventricle and right atrium, while patients are breathing room air and at end-expiration.
* Exercise capacity by means of a maximal incremental cycle testing (CardioPulmonary Exercise Test) to measure maximal work load, VO2 max, anaerobic threshold, heart rate response, oxygen pulse and ventilatory efficiency. And by means of 6 minute walking distance.
* Heart Rate Variability (HRV)
* Nuclear scanning: a comprised PET protocol will be performed to measure 11C-acetaat, oxygen-15-labeled water (H215O) and ¹¹C-HED uptake in the right ventricle. A summary of the protocol is added as a supplement.

UP-TITRATION PHASE (first 4 months; either on placebo or Bisoprolol): patients will be monitored every second week under supervision of an experienced pulmonologist, specialized in PAH, and a cardiologist, specialized in chronic heart failure during a visit to the outpatient clinic. If no contra-indications are found the dose will be increased to the next step.

The investigators will start with a dosage of 1,25 mg Bisoprolol once daily. Every two weeks dosage is increased by 1,25 mg, until maximum dosage of 10 mg once a day is reached, or as high as tolerated by the patient.

Increasing the dosage will be stopped, or if needed the dosage will be reduced, in case of:

* systolic systemic pressure < 90 mmHg
* clinical progression in heart failure
* clinically relevant bradycardia or <60b/min
* progression of complaints
* drop in 6 minute walk distance > 15% The titration procedure for the placebo will be the same as for titration of Bisoprolol. The dosage of the medication will be altered for maximal four months and after this the patients will use a stable dose for the rest of the six month period.

Every clinical visit will at least contain a clinical assessment, assessment of NYHA class, 6 minute walk distance, ECG and a Minnesota quality of life questionnaire. Every fourth week NT-proBNP, kidney- and liver functions will be assessed. In addition, the patient will be instructed to use a diary to record his/her symptoms and body weight.

STABLE PHASE: It is expected that up to 4 months are required to reach an acceptable dose of Bisoprolol. After this up-titration phase, the patient will be followed closely during the remaining part of the six month period, using a stable medication dose. The monitoring includes continuation of the diary, monthly visits to the outpatient clinic including the measurements as described in the up-titration phase and a telephone call every 4 weeks in between office visits.

CROSS OVER After six months new measurements will be done. Thereafter the medication will be tapered down in a two week period and than finally stopped. This will be done to prevent the patients for possible side effects (rebound tachycardia) of stopping their medication. The same tapering down procedure will be performed after the third set of measurements.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic PAH patients
* Stable on PAH specific treatment defined

  * No change in PAH specific treatment in the past 6 months
  * No change in functional class in the past 6 months
  * <10 % change in 6 minute walk distance in the past 6 months
* Functional class 2 or 3
* In sinus rhythm

Exclusion Criteria:

* History of systemic hypertension, ischaemic heart disease, valvular disease or cardiomyopathy.
* Asthma
* Use of concomitant medication other than diuretics, Acenocoumarol and PAH targeted therapy
* History of cardiac arrhythmias or the use of anti-arrhythmic drugs
* Sick sinus syndrome
* systolic hypotension < 90 mmHg
* AV-block
* Clinically relevant sinus-bradycardia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-02; Primary Completion 2014-01 (Actual); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Effectivity | 6 months
  The primary efficacy endpoint is improvement in RV function as reflected by RVEF determined by means of cardiac MRI.
Safety | continue
  Safety of Bisoprolol treatment in iPAH patients is not taken as a primary endpoint but seen as a precondition for this study and will be closely monitored. Dose titration will be guided by possible side effects.

SECONDARY OUTCOMES:
Is Bisoprolol treatment effective in reducing sympathetic overdrive? | 0,6,12 months
  Herefore the investigators use a C11-Hed-, H2O15- and a C11-acetate- nuclear scan
Is Bisoprolol effective in reversing maladaptive remodeling of the right ventricular wall, and does Bisoprolol thereby improve the diastolic properties of the right ventricle? | 0,6 and 12 months
  Pressure-Volume loops will be reconstructed from the combined right heart catheterization data and MRI measurements
Is Bisoprolol treatment effective in improving the perfusion and mechanical efficiency (oxygen consumption per joule) of the heart? | 0,6,12 months
  Perfusion will be measured by using the H2O tracer. Oxygen consumption of the right ventricle will be estimated from the uptake of the acetate tracer. Right ventricular power output will be derived from the right heart catheterization data.
Is Bisoprolol effective in improving exercise capacity? | Every two weeks
  This will be measured by means of the maximal oxygen uptake which is measured by means of the incremental cardiopulmonary exercise test and six minute walking distance.

CONTACTS AND LOCATIONS:
Overall Officials: Anton Vonk Noordegraaf, Prof. MD PhD, Principal Investigator — VU University Medical Center, pulmonary department
Locations (1):
- VUmc, Amsterdam, Netherlands

REFERENCES:
- [Derived] van Campen JS, de Boer K, van de Veerdonk MC, van der Bruggen CE, Allaart CP, Raijmakers PG, Heymans MW, Marcus JT, Harms HJ, Handoko ML, de Man FS, Vonk Noordegraaf A, Bogaard HJ. Bisoprolol in idiopathic pulmonary arterial hypertension: an explorative study. Eur Respir J. 2016 Sep;48(3):787-96. doi: 10.1183/13993003.00090-2016. Epub 2016 Jul 7. PMID 27390285